CLINICAL TRIAL: NCT02622386
Title: The Effect of Riboflavin on Moderate to Severe Plaque Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Johann E Gudjonsson MD PhD, Assistant Professor of Dermatology, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00105691 /Derm 677
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Riboflavin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riboflavin then Placebo (Experimental): Riboflavin (Vitamin B2) 400 mg oral capsule taken once daily for 12 weeks, followed by 4 week washout period before crossover. At crossover, patients will no longer receive Riboflavin but matching placebo capsule for additional 12 weeks.
  Interventions: Drug: Riboflavin
- Placebo then Riboflavin (Placebo Comparator): Placebo oral capsule taken once daily for 12 weeks, followed by 4 week washout period before crossover. At crossover, patients will no longer receive placebo but 400 mg Riboflavin (Vitamin B2) capsule for additional 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Riboflavin — Riboflavin (Vitamin B2) 400 mg capsule taken daily for 12 weeks.
  Other Names: Vitamin B2
  Arms: Riboflavin then Placebo
Other: Placebo — Matching placebo capsule taken daily for 12 weeks.
  Arms: Placebo then Riboflavin

SUMMARY:
The purpose of this study is to determine the anti-inflammatory effect of high-dose riboflavin supplementation on chronic plaque psoriasis. Psoriasis is a common chronic skin disorder that affects over 4 million people. There is no cure for psoriasis and treatment is directed at controlling patients' symptoms. Amongst patients with skin disease, there is significant interest in using complementary alternative medicine and vitamins to treat their disease. Previous human case reports suggest that riboflavin, commonly known as Vitamin B2, is clinically effective for the treatment of psoriasis; however, they were not conclusive. More recent human trials have shown that 400 mg of daily oral riboflavin is a safe and well-tolerated medication to administer to humans. For the purpose of this study, the riboflavin is used as an investigational drug.

DETAILED DESCRIPTION:
The purpose of this investigation is to determine the anti-inflammatory effect of high-dose riboflavin supplementation on chronic plaque psoriasis. Up to fifty volunteers with chronic plaque psoriasis will be recruited for a double-blind, placebo-controlled 28 week prospective study with cross-over of both the intervention and control groups at the 12 week time mark. There will be a 4 week washout period when subjects crossover. Riboflavin will be dosed 400 mg by mouth daily versus placebo. Throughout the study the investigators will perform both clinical and laboratory assessments to measure response.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Good general health
* Willingness and ability to follow the protocol
* Signed Informed Consent Form, written and witnessed.
* Stable moderate to severe chronic plaque psoriasis involving 8% or greater total body surface area (TBSA).
* If subject is a woman of childbearing potential, she must have a negative pregnancy test at screening and agree to use a medically acceptable form of contraception during the screening and throughout the study.

Exclusion Criteria:

* Started using a topical steroid stronger than moderate strength, vitamin A or D analog preparations, or anthralin within 14 days of study drug initiation.
* Initiated a systemic medications, including biologic medication, or phototherapy within 180 days of study drug initiation.
* Prior or concurrent use of cyclophosphamide.
* Currently using sulfasalazine therapy.
* Known hypersensitivity to riboflavin.
* Enrolled in any other investigational device or investigational drug trial(s) or receipt of any other investigational agent(s) within 28 days of baseline visit.
* Presence of severe comorbidities such as, diabetes mellitus requiring insulin; congestive heart failure (CHF) of any severity or myocardial infarction or cerebrovascular accident or transient ischemic attack within 3 months of screening visit; unstable angina pectoris, uncontrolled hypertension [sitting systolic BP <80 mm Hg or > 160 or diastolic BP > 100 mm Hg], oxygen-dependent severe pulmonary disease, history of cancer within 5 years [other than resected cutaneous basal or squamous cell carcinoma of the skin or in situ cervical cancer].
* Any of the following hematologic abnormalities, confirmed by repeat test at least 1 week apart:

  1. White blood count <3,000/µL or >14,000/µL
  2. Lymphocyte count <1,000/µL
  3. Neutrophil count <1,5000/µL
  4. Platelet count <150,000/µL
  5. Hemoglobin<10 g/dL
* Liver function test aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase (AlkP) results that are greater than or equal to 2 times the upper limit of normal (ULN).
* Serum creatinine ≥ to 2x the ULN.
* Known HIV-positive status or known history of any other immune-suppressing disease.
* Any current or past history of psychiatric disease that would interfere with ability to comply with study protocol or give informed consent.
* Had grade 3 or 4 adverse events or infections within 28 days before screening, or between screening visit and drug initiation.
* Evidence of any skin conditions other than psoriasis that would interfere with the evaluations of the effect of study medication on psoriasis.
* Presence of any condition or circumstances judged by the patient's physician, the investigator, or medically qualified study staff to render this clinical trial detrimental or otherwise unsuitable for the patient's participation.
* A history of non-compliance with other therapies.
* Females who are pregnant, lactating, planning on pregnancy during the study period, or unwilling to use FDA-approved method of birth control.
* A history of keloids or excessive scar formation or of healing poorly.
* A history of allergic reaction to local anesthetics, including lidocaine and epinephrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johann Gudjonsson, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Riboflavin Then Placebo: Riboflavin (Vitamin B2) 400 mg oral capsule taken once daily for 12 weeks, followed by 4 week washout period before crossover. At crossover, patients no longer received Riboflavin but matching placebo capsule for additional 12 weeks.
  Riboflavin: Riboflavin (Vitamin B2) 400 mg capsule taken daily for 12 weeks.
- Placebo Then Riboflavin: Placebo oral capsule taken once daily for 12 weeks, followed by 4 week washout period before crossover. At crossover, patients no longer received placebo but 400 mg Riboflavin (Vitamin B2) capsule for additional 12 weeks.
  Placebo: Matching placebo capsule taken daily for 12 weeks.
Period: First Assignment
Arm/Group | Riboflavin Then Placebo | Placebo Then Riboflavin
Started | 12 | 11
Completed | 9 | 9
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2
Period: Washout
Arm/Group | Riboflavin Then Placebo | Placebo Then Riboflavin
Started | 9 | 9
Completed | 5 | 5
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 4
Period: Second Assignment
Arm/Group | Riboflavin Then Placebo | Placebo Then Riboflavin
Started | 5 | 5
Completed | 5 | 3
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Because this is a crossover study, all Participants' data is combined.
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Customized [Count of Participants; unit: Participants]
  22 - 29 Years of Age | 1
  30 - 39 Years of Age | 0
  40 - 49 Years of Age | 8
  50 - 59 Years of Age | 8
  60 - 69 Years of Age | 5
  70 - 79 Years of Age | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
Psoriasis Area and Severity Index (PASI) at Baseline [Mean (Full Range); unit: score on a scale] — The range of absolute PASI scores is 0-72, with higher scores indicating a greater severity of psoriasis. 0 to <5=Mild psoriasis; 5 to <10 = Moderate psoriasis; 10 to <72 = Severe psoriasis.
  score on a scale | 8.7 [4.4 to 13.8]

OUTCOME MEASURES:

1. Primary Outcome: Subjects Achieving 50% or Greater Psoriasis Area and Severity Index (PASI) Reduction
Description: The number of subjects that achieve a 50 percent or greater reduction in their PASI with intervention as compared to placebo.
  The range of absolute PASI scores is 0-72, with higher scores indicating a greater severity of psoriasis. 0 to <5=Mild psoriasis; 5 to <10 = Moderate psoriasis; 10 to <72 = Severe psoriasis.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Riboflavin: Riboflavin (Vitamin B2) 400 mg oral capsule taken once daily for 12 weeks either before or after a 4-week washout period.
  Riboflavin: Riboflavin (Vitamin B2) 400 mg capsule taken daily for 12 weeks.
- Placebo: Placebo oral capsule taken once daily for 12 weeks either before or after a 4-week washout period.
  Placebo: Matching placebo capsule taken daily for 12 weeks.
Arm/Group | Riboflavin | Placebo
Number analyzed (Participants) | 17 | 16
Participants | 2 | 2

2. Secondary Outcome: Subjects Achieving PASI 75, 90, 100 Response
Description: The number of subjects that achieve a PASI 75, 90, 100 response with intervention as compared to placebo.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Riboflavin | Placebo
Number analyzed (Participants) | 17 | 16
Participants
  PASI 75 | 0 | 0
  PASI 90 | 0 | 0
  PASI 100 | 0 | 0

3. Secondary Outcome: Subjects Achieving Physician Global Assessment (PGA) Score 0/1
Description: The number of subjects that achieve a PGA score of 0/1 with intervention as compared to placebo. The Global Assessment Scale is a simple instrument with a 9 point ordinal scoring system ranging from -4 indicating very marked worsening to +4 very marked improvement. This scale provides a subjective overall evaluation of treatment response by the patients/caregivers or physicians/health care providers.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Riboflavin | Placebo
Number analyzed (Participants) | 17 | 16
Participants | 2 | 1

4. Secondary Outcome: Subjects Reporting Pruritus Score 0/1
Description: The number of subjects that report a pruritus score of 0/1 with intervention as compared to placebo. The pruritis scores can range from 0 to 10; where 0 means no itching and 10 means the worst itching.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Riboflavin | Placebo
Number analyzed (Participants) | 17 | 16
Participants | 0 | 2

5. Secondary Outcome: Subjects Reporting Dermatology Life Quality Index (DLQI) Score 0/1
Description: The number of subjects treated that report a DLQI score of 0/1 with intervention as compared to placebo. Minimum score 0, maximum score of 30, where 0 means dermatological problems are not causing impairment on their quality of life and 30 means extreme negative impact of dermatological conditions.
  0-1 = no effect at all on patient's life; 2-5 = small effect on patient's life; 6-10 = moderate effect on patient's life; 11-20 = very large effect on patient's life; 21-30 = extremely large effect on patient's life.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Riboflavin | Placebo
Number analyzed (Participants) | 17 | 16
Participants | 2 | 3

6. Secondary Outcome: Difference in Riboflavin Serum Plasma Levels and Flavin-adenine Dinucleotide (FAD)
Description: The difference in serum plasma levels of riboflavin and FAD in subjects treated with intervention as compared to placebo.
Time Frame: 12 weeks
Population: Not available as assays were not able to be conducted.
Arm/Group | Riboflavin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were followed for 32 weeks (12 weeks of treatment 1; 4 weeks of washout; 12 weeks of treatment 2; and 4 weeks of followup)
Arm/Group | Riboflavin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 9/17 | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riboflavin (N=17) | Placebo (N=16)
sinus infection (Infections and infestations) | 1 | 1
acid reflux flare (Gastrointestinal disorders) | 0 | 1
elevated liver enzymes (Hepatobiliary disorders) | 1 | 0
elevated blood pressure (Cardiac disorders) | 1 | 0
fatigue (General disorders) | 1 | 1
worsening psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
biopsy reaction (General disorders) | 1 | 1
migraine aura (Nervous system disorders) | 1 | 0
abdominal plasty (Surgical and medical procedures) | 1 | 0
allergies (General disorders) | 0 | 2
cold (Infections and infestations) | 1 | 1
24 hour Gastrointestinal event (Infections and infestations) | 0 | 1
upper respiratory infection (Infections and infestations) | 1 | 0
eye itching (Eye disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 0 | 1
flu (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT02622386/Prot_SAP_000.pdf